CLINICAL TRIAL: NCT02911714
Title: A Pilot Study to Develop Contrast-Enhanced Ultrasound for Kidney Transplant
Brief Title: Contrast-Enhanced Ultrasound for Kidney Transplant
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: lack of funding
Sponsor: University of Utah (Other)
Collaborators: National Kidney Foundation, United States (Other); American Heart Association (Other); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB_00092223; KL2TR002539 (NIH)
Record Dates: First submitted 2016-09-19; First posted 2016-09-22 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Kidney Transplantation
Keywords: Kidney Transplantation; Delayed Graft Function; Acute Allograft Rejection; Acute Kidney Injury
MeSH Terms: conditions — Delayed Graft Function; Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CEUS and Delayed Graft Function (Experimental): On the first post-operative day after kidney transplantation, recipients enrolled in the study will undergo CEUS using Lumason to quantify microvascular perfusion within the cortical and medullary zones of the kidney allograft for comparison to the concentration of neutrophil gelatinase-associated lipocalin (NGAL, an early biomarker of acute kidney injury) measured from recipient urine simultaneously collected on the first post-operative day.
  Interventions: Drug: Lumason Contrast-Enhanced Ultrasound
- CEUS and Biopsy-Proven Acute Rejection (Experimental): We will identify and enroll kidney transplant recipients in need of clinically-indicated duplex ultrasounds and possible biopsy to evaluate allograft dysfunction during hospital admissions and outpatient follow-up. Immediately after the duplex ultrasound, we will perform CEUS using Lumason for allograft perfusion measurements to determine its potential association with biopsy-proven acute rejection according to the most recent Banff criteria.
  Interventions: Drug: Lumason Contrast-Enhanced Ultrasound

INTERVENTIONS:
Drug: Lumason Contrast-Enhanced Ultrasound — In both arms, we will use Lumason to measure kidney allograft perfusion via contrast-enhanced ultrasound.
  Other Names: Sulfur hexafluoride lipid-type A microspheres

SUMMARY:
Contrast-enhanced ultrasound (CEUS) is a promising non-invasive imaging tool that may aid in the early detection of kidney transplant complications, such as delayed graft function (DGF) and acute allograft rejection. The technique uses an intravenous contrast agent to improve organ visualization with standard duplex ultrasound equipment. A number of FDA-approved agents, including Optison, Definity and Lumason are widely used to improve visualization in technically limited echocardiograms, and Lumason was recently approved for contrast-enhanced ultrasound of the liver. The specific aims of this study are to: develop, implement and refine a contrast-enhanced ultrasound protocol using Lumason to safely maximize kidney allograft visualization; determine associations between contrast-enhanced ultrasound and patterns of allograft injury consistent with delayed graft function; and to compare contrast-enhanced ultrasound with duplex ultrasound for differentiating acute rejection from other causes of dysfunction.

DETAILED DESCRIPTION:
Kidney transplantation is the preferred treatment for end-stage renal disease (ESRD) given improved quality of life, longer survival and lower costs compared with chronic dialysis. Despite these long-term benefits, the first year post-transplant is a critical period that influences health care costs for transplantation and long-term patient and allograft survival. The two most common complications in the first year are delayed graft function (DGF), which affects nearly 25% of deceased-donor transplants, and acute allograft rejection, which affects nearly 10% of all transplants (deceased and living donor). DGF is most commonly caused by severe ischemia-reperfusion injury at transplantation and is a known risk factor for acute rejection and premature failure. Driven by an ever-growing transplant waiting list and limited organs, efforts to utilize higher-risk kidneys for increasingly higher-risk recipients may further increase these complication rates. While treatments exist for DGF and acute rejection, the current diagnostic paradigm is to obtain a duplex ultrasound (DUS) of the allograft, based on serial changes in serum creatinine, and then proceed to biopsy if there is clinical concern for rejection. Biopsy is the gold standard to differentiate between causes of allograft dysfunction, but the procedure is invasive and typically takes 24 hours or longer for an interpretation. Thus, early detection of these complications using non-invasive diagnostic methods (a major transplant research goal) could reduce our reliance on biopsies and help improve long-term patient and allograft survival.

Researchers in the United States have safely performed contrast-enhanced ultrasounds of the kidney in healthy participants, and radiologists have used ultrasound contrast agents off-label to better visualize organs other than the heart when clinically indicated. In terms of kidney transplants, European data suggest CEUS of the allograft on post-operative day (POD) 7 is superior to DUS for predicting 12-month allograft function, but there are no published studies using CEUS on POD 1 to diagnose DGF or acute rejection.

The pathophysiology of both DGF and acute rejection involve interactions between the microvasculature, parenchymal cells and inflammatory cells, though with differences in timing and within different zones of the kidney itself. A very important feature of CEUS is its capacity to measure microvascular perfusion, whereas DUS can only estimate flow within larger vessels. This potential innovation for assessing the renal macro- and microvasculature may allow for earlier non-invasive detection of DGF and acute rejection. With additional research, it may ultimately be shown that non-invasive CEUS will revolutionize early DGF and acute rejection diagnosis to enable improvement in long-term patient and allograft survival.

ELIGIBILITY:
Inclusion Criteria:

* Adult living-donor or deceased-donor kidney transplant recipients

Exclusion Criteria:

* Subject is Pregnant
* History of non-renal transplant
* Uncontrolled diabetes or hypertension
* Symptomatic or significant pulmonary or cardiovascular disease
* Clinical decision by the treating team to forego the study procedure due to medical/surgical instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Biomarker-Defined Delayed Graft Function | Post-Operative Day 1
  A meta-analysis of 19 studies found urine neutrophil gelatinase-associated lipocalin (NGAL) >150 ng/mL (within hours of the inciting event) had an area under the receiver-operating characteristic curve (AUC) of 0.815 for identifying acute kidney injury (defined as an ensuing rise in serum creatinine by ≥50%). We noted an AUC of 0.82 for predicting the need for dialysis in the first week (i.e., dialysis-defined delayed graft function) with an optimal urine NGAL cutoff of >350 ng/mL. For this study outcome, we will determine the Spearman correlation between CEUS-assessed allograft perfusion and degree of allograft injury based on post-operative day 1 urine NGAL concentration.
Biopsy-Proven Acute Rejection | Any Time After Kidney Transplantation
  The Banff (2013) classification of acute kidney allograft rejection requires histologic evidence of acute tissue injury, evidence of recent antibody interaction with renal vascular endothelium, and serologic evidence of donor-specific antibodies in order to diagnose acute antibody-mediate rejection. Acute T-cell mediated rejection is histologically graded by the extent of interstitial inflammation and vascular involvement.

SECONDARY OUTCOMES:
Dialysis-Defined Delayed Graft Function | First Post-Operative Week
  The need for any dialysis in the first week of transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Isaac E Hall, M.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah Hospital, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No